CLINICAL TRIAL: NCT02219334
Title: Comparing Nasal Suction Devices in Children With Bronchiolitis: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to low enrollment.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Shabana Yusuf, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-33659
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Bronchiolitis
Keywords: Children; Nasal suction devices; Suctioning
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NoseFrida (Experimental): If randomized to the NoseFrida group, the NoseFrida/filters will be given along with educational instruction of its use to the parents of patients admitted with bronchiolitis. The NoseFrida will be used by the parent to suction the nares of their infants/toddlers.
  Interventions: Device: NoseFrida
- NeoSucker (No Intervention): The NeoSucker (used for nasal suctioning) is part of the current standard of care for patients with bronchiolitis. The NeoSucker is used for removing nasal secretions by a nurse or respiratory therapist. The NeoSucker is a plastic tube which is used to suction the secretions. The bedside nurse will continue to use the NeoSucker as needed. NoseFrida will not be used for this sub group of patients.

INTERVENTIONS:
Device: NoseFrida — The NoseFrida has four components, the collection container, an interchangeable filter, flexible tubing and a mouth piece. The end of the collection devise is placed on the patient's nostril, a tight seal is made via the vacuum created from suctioning of the mouth piece and secretions are easily aspirated. This device disassembles for quick disinfecting and cleaning.
  Arms: NoseFrida

SUMMARY:
The purpose of our study is to determine the safety, efficacy, length of stay and parental satisfaction of the NoseFrida in comparison to a suction device used in the hospital setting in patients with bronchiolitis admitted under observation status.

DETAILED DESCRIPTION:
Bronchiolitis is a viral illness and a common cause for admission to the hospital. Most patients with bronchiolitis are managed at home. The indications of hospitalization are poor feeding (due to increased mucus production) and respiratory distress with and without hypoxia. The acute care setting is a common destination of patients with bronchiolitis. Patients are admitted to the acute care setting for respiratory monitoring, suctioning and poor oral intake. The management of bronchiolitis is mostly supportive which includes frequent feedings, nasal suctioning, intravenous fluids and oxygen if necessary. The patients admitted to the acute care setting receive frequent nasal suctioning by a suction device (NeoSucker) and deep suctioning as needed. Since young infants are "nose breathers," the use of nasal suctioning helps to relieve nasal congestion/upper airway obstruction and assists with their ability to breathe and feed. Suctioning can be accomplished by the use of the bulb suction, nasal aspirators and/or suction catheters connected to pressure devices.

The role of the type of suctioning device in the management of bronchiolitis has not been studied extensively. In our study, a nasal aspirator (developed in Sweden by an Ear, Nose and Throat specialist) by the brand name of NoseFrida will be compared to the NeoSucker, a suction catheter currently used in our hospital setting which requires both a nurse and a pressure device. Nasal suctioning is less traumatic and does not cause the discomfort, bleeding and rebound swelling that deep suctioning can. Upon admission, patients will be randomized to either the NoseFrida or NeoSucker group. After consent is obtained for agreed participation, the patients parents randomized to the NoseFrida group will be given a NoseFrida/filters and instructions on usage (instructional video/postcard). The parents will be encouraged to use the NoseFrida suction device as often as they want, especially before feeds and sleep. The patients randomized to the NeoSucker group will be given the current standard of care and nasal suctioned by a nurse. Both groups will be deep suctioned as clinically needed.

ELIGIBILITY:
Inclusion Criteria:

* patients above the age of 2 months and post-gestational age to 44 weeks and less than or equal to 2 years with signs and symptoms of bronchiolitis
* clinical respiratory score (CRS) of less than or equal to 4
* principle diagnosis of bronchiolitis (International Classification of Diseases-9: 466, 466.11 and 466.19)
* Patient admitted to the Pediatric Hospitalist Medicine (PHM) group
* Patient with associated hypoxemia and/or respiratory distress requiring low flow O2 nasal cannula (NC) management (2L/min or less)

Exclusion Criteria:

* age less than 2 months
* age less than post-gestational age 44 weeks
* CRS greater than 4
* associated hypoxia
* already using NoseFrida at home
* chronic lung disease
* oro-facial abnormalities
* cardiac abnormalities

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth L Watson, MSN, RN, CNL, Study Director — Baylor College of Medicine; Aderonke Adekunle-Ojo, MD, Study Chair — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benincaso FV, Smith MH. A suction-controlled nasal aspirator for collection of nasopharyngeal secretions. J Pediatr. 1973 Feb;82(2):297-9. doi: 10.1016/s0022-3476(73)80175-1. No abstract available. PMID 4684375
- [Background] Budhiraja, S., Verma, R., Shields, M.D. (2012). The management of acute bronchiolitis in infants. Paidiatrics and Child Health, 23(7), 296-300.
- [Background] Casati M, Picca M, Marinello R, Quartarone G. Safety of use, efficacy and degree of parental satisfaction with the nasal aspirator Narhinel in the treatment of nasal congestion in babies. Minerva Pediatr. 2007 Aug;59(4):315-25. PMID 17947838
- [Background] Da Dalt L, Bressan S, Martinolli F, Perilongo G, Baraldi E. Treatment of bronchiolitis: state of the art. Early Hum Dev. 2013 Jun;89 Suppl 1:S31-6. doi: 10.1016/S0378-3782(13)70011-2. PMID 23809346
- [Background] Deshpande SA, Northern V. The clinical and health economic burden of respiratory syncytial virus disease among children under 2 years of age in a defined geographical area. Arch Dis Child. 2003 Dec;88(12):1065-9. doi: 10.1136/adc.88.12.1065. PMID 14670770
- [Background] Diagnosis and Managment of Bronchiolitis., 2006. Subcommittee on Diagnosis and Management of Bronchiolitis. 118, 1774.
- [Background] Hall CB, Weinberg GA, Iwane MK, Blumkin AK, Edwards KM, Staat MA, Auinger P, Griffin MR, Poehling KA, Erdman D, Grijalva CG, Zhu Y, Szilagyi P. The burden of respiratory syncytial virus infection in young children. N Engl J Med. 2009 Feb 5;360(6):588-98. doi: 10.1056/NEJMoa0804877. PMID 19196675
- [Background] Jarvis K, Pirvu D, Barbee K, Berg N, Meyer M, Gaulke L, Pate BM, Roberts C. Change to a standardized airway clearance protocol for children with bronchiolitis leads to improved care. J Pediatr Nurs. 2014 May-Jun;29(3):252-7. doi: 10.1016/j.pedn.2013.11.007. Epub 2013 Nov 27. PMID 24333327
- [Background] Moore T. Suctioning techniques for the removal of respiratory secretions. Nurs Stand. 2003 Nov 12-18;18(9):47-53; quiz 54-5. doi: 10.7748/ns2003.11.18.9.47.c3504. PMID 14649194
- [Background] Mussman GM, Parker MW, Statile A, Sucharew H, Brady PW. Suctioning and length of stay in infants hospitalized with bronchiolitis. JAMA Pediatr. 2013 May;167(5):414-21. doi: 10.1001/jamapediatrics.2013.36. PMID 23460088
- [Background] Nagakumar P, Doull I. Current therapy for bronchiolitis. Arch Dis Child. 2012 Sep;97(9):827-30. doi: 10.1136/archdischild-2011-301579. Epub 2012 Jun 25. PMID 22734014
- [Background] Sandweiss DR, Corneli HM, Kadish HA. Barriers to discharge from a 24-hour observation unit for children with bronchiolitis. Pediatr Emerg Care. 2010 Dec;26(12):892-6. doi: 10.1097/PEC.0b013e3181fe911d. PMID 21088635
- [Background] Wai AK, Kwok WO, Chan MS, Graham CA, Rainer TH. Patients' perceptions of nasopharyngeal aspiration in the emergency department of a teaching hospital in Hong Kong. Emerg Med J. 2007 Jan;24(1):35-6. doi: 10.1136/emj.2006.039701. PMID 17183041

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NoseFrida | NeoSucker
Started | 32 | 23
Completed | 24 | 20
Not Completed | 8 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NoseFrida | NeoSucker | Total
Number analyzed (Participants) | 24 | 20 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 20 | 44
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 14 | 13 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Length of stay [Median (Inter-Quartile Range); unit: Hours] | 26.23 [17.63 to 40.48] | 25.13 [19.70 to 45.42] | 25.93 [19.48 to 43.18]

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Median Length of Stay of the Two Devices in Hours
Description: The study group will analyze the length of stay for the NoseFrida group and compare it with the NeoSucker group.
Time Frame: Participants will be followed for the duration of their stay in the EDOU, up to 48 Hours or end of hospitalization whichever is greater
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | NoseFrida | NeoSucker
Number analyzed (Participants) | 24 | 20
Hours | 26.23 [17.63 to 40.48] | 25.13 [19.70 to 45.42]
Statistical Analysis 1: Comparison: NoseFrida vs NeoSucker; The primary hypothesis of length of stay equivalence within a margin of ± 5 hours was tested using the two one-sided t-test (TOST) procedure, with a 5% significance level; Test type: Equivalence — Historical data at the institution for similar patients had a mean length of stay(LOS) of 25.7 hours (standard deviation-[SD] =10.3) from 9/2012- 9/13 was observed for 134 patients admitted to the emergency department observation unit and treated with the standard of care (NeoSucker). Given a LOS-SD of 10.3 hours, 75 subjects per treatment group would provide 80% statistical power at the 5% significance level to demonstrate equivalence in the two treatments' length of stay within ±5 hours; p < 0.05, two one-sided t-test (TOST); Mean Difference (Final Values) = 2.49, 95% CI 2-sided [-10.74 to 15.72], Standard Deviation 21.4 — Due to slower than anticipated patient recruitment, the target size of 75 participants per treatment group was not reached

2. Other Pre Specified Outcome: Percentage of Patients Readmitted Within 48 Hours of Discharge.
Description: The study group will analyze those patients both from the NoseFrida group and the NeoSucker group who are readmitted within 48 hours of discharge from the EDOU.
Time Frame: within 48 hours of discharge
Measure: Count of Participants; unit: Participants
Arm/Group | NoseFrida | NeoSucker
Number analyzed (Participants) | 24 | 20
Participants | 1 | 0

3. Other Pre Specified Outcome: Parental Satisfaction (NoseFrida Group) Will be Measured Using a Newly Developed Survey Tool (Likert Scale).
Description: A study specific survey was developed to measure parental satisfaction of the NoseFrida device. The parental satisfaction question responses were on a 5 point Likert Scale as follows: 1="Strongly Disagree", 2="Disagree", 3="Neutral", 4="Agree" and 5="Strongly Agree." The minimum value is strongly disagree and maximum is strongly agree. The likert scale assessed parental satisfaction with the use of the device.
Time Frame: as for outcome 1
Population: Parental satisfaction survey was only done on Nosefrida group since the Neosucker is the standard of care
Measure: Median (Full Range); unit: score on a scale
Arm/Group | NoseFrida | NeoSucker
Number analyzed (Participants) | 24 | 0
score on a scale | 5 [1 to 5] |

ADVERSE EVENTS:
Time Frame: Adverse reaction was monitored throughout the hospital stay "an average of 26 hours" till the patient was discharged. No adverse event monitoring was done after discharge.
Arm/Group | NoseFrida | NeoSucker
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/23
Other Adverse Events (participants affected / at risk) | 0/32 | 0/23

LIMITATIONS AND CAVEATS:
The sample size was small and was a convenience sample. Not all parents participated in the satisfaction survey. The lack of documentation of nose bleeds and nasal swelling does not suggest the absence of these minor side effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT02219334/Prot_SAP_000.pdf